CLINICAL TRIAL: NCT07258342
Title: Evaluation of the Effects of Closed Kinetic Chain Exercises and Kinesio Taping on the Lower Extremity in Individuals With Chronic Stroke
Brief Title: Evaluation of Lower Extremity Interventions in Individuals With Chronic Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Sezen Pehlivan, Master's Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-SBF-FTR-01
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Chronic Stroke Patients; Lower Extremity; Knee Proprioception; Closed Kinetic Chain Exercises; Kinesiotape; Physiomaster

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group engaged in closed kinetic chain exercises (Experimental): Closed kinetic chain exercises of the lower extremity are typically performed with the feet secured to a stable object that generates compressive forces at the hip, knee, and ankle joints. Participants will perform closed kinetic chain exercises in 40-minute sessions, twice a week for 8 weeks. Each exercise will be repeated 3 to 5 times, depending on the individual's strength .Exercises include: wall squats, forward and upward step-ups, side and upward step-ups, double-leg squats, bridges, and quadriceps isometric strengthening exercises.
  Interventions: Other: Measurement of Knee Joint Position Sense; Other: Berg Balance Scale (BDS); Other: Timed Up and Go Test (TUG); Other: 10-Meter Walking Test; Other: Stroke-Specific Quality of Life Scale
- Kinesiotaping Group (KB) (Experimental): Kinesiotaping will be applied to increase proprioceptive awareness of the knee joint. Taping will be applied using the *"Y" technique and *"I" technique, focusing on medial and lateral support. The kinesio tape will remain in place for 3 days, followed by a 1-day break, and then reapplied. Tape changes will be performed by a physical therapist for a total of 8 weeks.
  Interventions: Other: Measurement of Knee Joint Position Sense; Other: Berg Balance Scale (BDS); Other: Timed Up and Go Test (TUG); Other: 10-Meter Walking Test; Other: Stroke-Specific Quality of Life Scale

INTERVENTIONS:
Other: Measurement of Knee Joint Position Sense — Joint position sense will be assessed using active and passive joint position sense tests. Before starting the movement, the extremity will be moved ten times to prepare for movement. The "Physio Master" phone application will be used to measure the angle difference between the affected and unaffected knees at the end point of the movement. With the individual sitting upright with their back straight, knees flexed at 90 degrees, the participant's knee will be flexed to 45 degrees and the participant will be asked to repeat the same angle with their eyes closed. The error in angles (°) will be calculated. Passive position sense will be measured and recorded by passively moving the participant to the determined angle (15-30-45-60) and then asking them to estimate the angle upon returning to the starting position. Repeated flexion and extension will be performed to assess any errors in the movement. Placebo exercises will also be administered during the assessment. The test was repeated t
Other: Berg Balance Scale (BDS) — The Berg Balance Scale was developed primarily to assess postural control and is widely used in many rehabilitation settings. The 14 items in the scale assess expected balance during common activities of daily living, including standing and static sitting balance, as well as turning, picking up objects from the floor, and transfers. Scoring is typically done on a 5-point scale that assesses whether the patient can perform the task safely and independently for a specific time period. A score of 0 is given when the patient cannot perform the movement at all, and a score of 4 is given when the patient completes the movement independently. The maximum score is 56, with a score of 0-20 indicating impaired balance, 21-40 indicating acceptable balance, and 41-56 indicating good balance. The completion of the scale takes approximately 10 to 20 minutes. The Turkish validity and reliability study of the scale was conducted by Şahin et al. in 2008 on stroke patients.
Other: Timed Up and Go Test (TUG) — It measures the time it takes for a patient to stand up from a chair, walk 3 meters, turn, and sit back down. The test time was recorded in seconds. The test was repeated three times, and the average time was recorded as a score. If necessary, the patient was allowed to perform the test using a walking aid. It is an objective clinical measurement used to assess functional mobility, dynamic balance, and fall risk in older individuals. It has also been shown to be a valid and reliable test in stroke patients.
Other: 10-Meter Walking Test — This test is used to determine walking speed. Two to three trials will be conducted at both comfortable and maximum speeds of their choosing. Participants will be instructed to walk at a "normal comfortable speed" or "as fast as safely possible." No practice trials will be conducted, and participants will rest for at least 30 seconds between trials. Typical shoes, standard orthotics, and any necessary assistive devices will be worn. Participants will walk approximately 14 meters, including a 2-meter acceleration and deceleration zone. The time participants spend walking the middle 6 meters of this walkway will be measured with a stopwatch, from the moment their toes first pass the starting cone to the moment they first pass the finishing cone. Walking speed will be calculated for each trial.
Other: Stroke-Specific Quality of Life Scale — Quality of life is also an important prognostic indicator for stroke and provides a broader definition of the disease. This scale consists of 49 items in 12 domains: mobility, energy, upper extremity functionality, work/productivity, mood, self-care, social roles, family roles, vision, language, thinking, and personality. SS-QOL items are assessed on a five-point Likert-type scale. Responses range from 1 (Strongly disagree) to 5 (Strongly agree). High scores on the scale indicate high quality of life, while low scores indicate low quality of life.

SUMMARY:
This study aims to evaluate the effectiveness of closed kinetic chain (CKC) exercises and kinesio taping on knee joint proprioception, balance, functional performance, and quality of life in individuals with chronic stroke. Stroke often results in proprioceptive deficits and postural control impairments, which negatively impact rehabilitation outcomes. While CKC exercises are believed to enhance proprioceptive input through joint compression and sensory feedback, kinesio taping is used as a complementary intervention to support motor control and stability. The study will compare the effects of these two interventions to determine their potential roles in improving sensorimotor function and promoting functional independence in stroke rehabilitation.

A total of 30 participants were enrolled in this study.

Inclusion Criteria:

* Patients who had a stroke more than 6 months ago,
* Having a stable medical condition,
* Ability to understand simple instructions,
* Individuals with spasticity between grades 0-2 according to the Modified Ashworth Scale,
* Individuals who can walk independently or with assistive devices,
* Those who agree to participate and comply with the study procedures.

Exclusion Criteria:

* Severe cognitive impairment (MMSE score < 24),
* Orthopedic conditions that may cause knee pain during exercise,
* Other neurological conditions that may affect proprioception,
* Severe joint contracture,
* Refusal or unwillingness to participate in the study.

DETAILED DESCRIPTION:
Stroke is defined as a sudden loss of neurological function lasting more than 24 hours, occurring in central nervous system regions such as the brain, spinal cord, or retina, due to infarction or hemorrhage. Etiologically, stroke is classified into two main groups: hemorrhagic and ischemic. Ischemic stroke occurs due to insufficient blood flow to cerebral tissue, while hemorrhagic stroke is characterized by bleeding into brain tissue or the subarachnoid space. Of all stroke cases, approximately 44% occur in men and 56% in women. The prevalence of stroke is around 22% in individuals aged 15 to 49 and increases to 67% when examined up to the age of 70.

The post-stroke period is typically divided into phases. The Stroke Roundtable Consortium recommends the following classification: the first 24 hours as the hyperacute phase, the first 7 days as the acute phase, the first 3 months as the early subacute phase, months 4 to 6 as the late subacute phase, and after 6 months as the chronic phase.

Following a stroke, patients commonly experience postural control loss, asymmetric weight distribution, abnormal gait patterns, and balance impairments, all of which negatively affect functional independence and quality of life.

Sensory deficits are also prevalent in stroke patients, with exteroception affected in 7-53%, proprioception in 34-64%, and higher cortical functions in 31-89% of cases. Most patients experience impairments in multiple types of sensation. These sensory disturbances reduce the feedback received from objects, potentially leading to non-use of the affected limb. Among these, proprioceptive deficits pose significant challenges during rehabilitation. Studies have shown that reduced proprioception in individuals with stroke negatively affects motor control and should be addressed in rehabilitation programs.

Progressive resistance exercise has been shown to be an effective treatment for strengthening weak muscles caused by various musculoskeletal and neuromuscular disorders. It is a training method that gradually increases the level of resistance to improve force generation capacity. Closed kinetic chain (CKC) and open kinetic chain (OKC) exercises are two widely used progressive resistance training methods aimed at improving proprioception and motor functions in stroke patients. CKC exercises are believed to enhance proprioception by providing greater sensory feedback through joint position sense and mechanoreceptor activation.

CKC exercises are typically performed with the terminal segment of a limb fixed and in continuous contact with a surface, resulting in compressive forces through the joints of the lower extremities. In contrast, OKC exercises are performed with the terminal segment of the limb free to move and are reported to primarily increase muscle strength rather than improve proprioception during movements like knee flexion and extension. Previous studies suggest that CKC exercises may offer more sensory input, thereby enhancing sensorimotor functions, including motor control and joint proprioception, more effectively than OKC exercises.

Kinesio taping, a method that can improve function in stroke patients, is used as a complementary treatment due to its positive effects on postural control, muscle strength, mobility, balance, and gait patterns. However, most previous studies have focused on ankle joint applications of kinesio taping, and only a limited number have examined its effects on proprioception, postural control, and gait when combined with proprioceptive training targeting the knee joint in stroke patients.

Proprioceptive training, as a method that enhances proprioception in stroke patients, is mainly utilized to determine the effectiveness of new rehabilitation approaches.

The aim of this study is to evaluate knee joint position sense in individuals with chronic stroke and to comparatively examine the effectiveness of closed kinetic chain exercises and kinesio taping in improving this sense. The study aims to assess the effects of these two interventions on proprioception, balance, functional performance, and quality of life.

The post-stroke recovery process, while individual differences persist, is examined in three main phases: acute, subacute, and chronic. The chronic stroke phase is generally defined as the period six months or more after the stroke and is the phase in which the patient's functional status stabilizes. However, the potential for recovery continues during this phase with neuroplasticity and rehabilitation interventions.

Neurological recovery (Neuroplasticity) refers to the structural and functional reorganization of the brain. Neuroplasticity occurs as an adaptive response to brain damage. This process involves the restructuring of nerve cells, glial cells, and axons. These mechanisms are most intense in the early stages of post-stroke recovery, especially in the first six months (88).

Recovery from stroke occurs through mechanisms such as neuroplasticity, the reorganization of adjacent brain regions, the strengthening of synaptic connections, and the activation of alternative neural pathways (89).

Functional recovery refers to individuals becoming more independent in their daily activities. Post-stroke recovery generally begins rapidly in the first six months and shows significant improvement within a year (90). Functional recovery depends not only on neurological recovery but also on the environmental and psychological interactions of patients. Patients typically experience a decrease in muscle tone (flaccid phase) initially after a stroke. However, this phase typically gives way to a spastic phase with increased muscle tone. This transition begins within 2-4 weeks. A prolonged flaccid phase and a late onset of tone increase indicate a poor recovery prognosis. Furthermore, delayed return of reflexes, excessive proximal muscle tone, and the absence of voluntary hand movement negatively impact the expectation of functional recovery (88). Post-stroke recovery generally progresses from proximal to distal, with the highest potential for recovery within the first 6 months. During this period, 80% of individuals require rehabilitation, 10% do not benefit from treatment, and another 10% may recover spontaneously (91).

Many factors influence recovery and functional outcomes:

* Stroke location and size: Cortical strokes generally have a worse prognosis than subcortical strokes (92).
* Early motor function status: Motor function level in the first weeks is the strongest predictor of long-term functional recovery (93).
* Age: Younger patients have a higher potential for recovery (94).
* Cognitive and psychosocial status: Depression, lack of motivation, and cognitive impairments negatively impact rehabilitation success (95).

4.10 The Importance of Physiotherapy and Rehabilitation in Chronic Stroke During this period, the patient may have regained much of the movement lost due to the stroke. Tone may be approaching normal, but significant deficits in timing and coordination skills are evident. Physical therapy goals are the cornerstone of stroke rehabilitation, encompassing a multifaceted approach aimed at restoring mobility, improving motor function, and alleviating physical impairments. The goals include restoring normal walking and stair activities, improving manual dexterity and grasping abilities, and improving cardiorespiratory endurance. (96,97) Stroke treatment begins with the patient's clinical condition stabilizing. Early intervention helps preserve brain tissue and supports the penumbra. It also prevents learned disuse and compensatory strategies, allowing the neuroplasticity process to progress properly (98). In the acute phase, it is important to protect the patient from complications. During this period, the goal is to prevent potential complications such as pneumonia, deep vein thrombosis, pulmonary embolism, and cardiac arrhythmias. Early mobilization, in-bed exercises, positioning, and cardiopulmonary rehabilitation approaches support the patient's functional recovery. For patients transitioning to the subacute phase, more advanced rehabilitation methods are implemented. During this period, exercises aimed at improving mobility, balance, sitting training, and upper extremity function and sensory integration are implemented. At the same time, treatment continues in parallel with areas such as occupational therapy, speech and language therapy, swallowing rehabilitation, and cognitive rehabilitation.

In the chronic phase, comprehensive rehabilitation approaches tailored to the patient's needs continue through inter- and multidisciplinary teamwork and home programs. Any existing complications are treated (47). Therapists use various balance exercises and proprioceptive activities to improve the balance and coordination necessary to prevent falls and maintain functional mobility. These exercises generally involve challenging the patient's balance in a controlled environment to improve balance reactions and postural control (99).To reduce the risk of secondary complications such as joint contractures and stiffness, therapists incorporate range-of-motion exercises. These exercises aim to maintain joint flexibility, prevent musculoskeletal problems, and facilitate range of motion in the affected limbs (91,100). They extend beyond clinical settings to include functional training and home modification recommendations. The therapist collaborates with patients to simulate activities important to daily living through practice. Additionally, they provide guidance on adapting their home environment and recommend assistive devices and modifications to improve accessibility and safety in the home environment. (101,102) 4.11 Physiotherapy Rehabilitation Approaches in Chronic Stroke Rehabilitation interventions in the chronic phase generally include community-based programs that provide ongoing therapy and support. PNF patterns and repetitive contractions can be used. Controlled eccentric contractions are necessary to restore normal function. Protective extension reactions should be introduced. (103) Balance and gait training should be performed at different speeds and difficulties. Advanced therapies such as robot-assisted therapy and virtual reality training are used to improve motor skills and cognitive functions. Biofeedback can be used to prompt the patient to perform voluntary muscle contractions in weak muscles. (104,105) Functional electrical stimulation (FES) can be used to improve muscle function, and mirror therapy can be used to create the illusion of movement in the affected limb. (106) Cognitive rehabilitation activities are designed to improve memory, attention, and problem-solving skills. Aerobic exercises and hydrotherapy are included to improve cardiovascular health and overall fitness (71). Music therapy can be beneficial for improving mood and cognitive function (107). Long-term psychological support is crucial for helping patients adapt to their new normal and maintain their motivation to continue their recovery (108).

Methods applied in stroke rehabilitation can be categorized as neurophysiological approaches, conventional treatments, and functional treatments.

Among neurophysiological approaches, the Proprioceptive Neuromuscular Facilitation (PNF) technique, which aims to improve motor control and muscle function by facilitating and relearning motor responses through proprioceptive stimulation, is one of the most popular. The Bobath approach, which utilizes the brain's neuroplasticity to reduce abnormal movement patterns and support the regaining of normal motor functions, is among the most popular approaches. Additionally, the Brunnstrom method and the Johnstone and Rood approach are also among the neurophysiological approaches.

Conventional treatments include range of motion, strengthening and stretching exercises, balance and coordination and gait training, thermotherapy methods, electrotherapy agents, orthotic approaches, manual therapy techniques, and mat exercises.

Functional approaches, on the other hand, include various technological approaches such as mirror therapy, forced restraint therapy and biofeedback, virtual reality applications, and robot-assisted rehabilitation. (48,109,110) 4.12 Sensory Impairment in Chronic Stroke Stroke is a sudden and focal lesion of the central nervous system and usually results from occlusion or hemorrhage in cerebral vessels. In the post-stroke period, in addition to motor function losses, significant impairments in the sensory system are observed. These sensory system impairments severely limit patients' ability to maintain activities of daily living and create significant challenges in the rehabilitation process. (111) The Role of the Sensory System in Stroke: The primary functions of the sensory system include superficial sensations such as touch, pain, and temperature, as well as deep sensations such as proprioception and vibration. Depending on the location of the stroke lesion, damage to any or more of these senses may occur. Proprioceptive impairments, in particular, are critical for motor control because knowing the position of muscles and joints is essential for coordination and balance (8).

Studies in chronic stroke patients have shown that the rate of superficial and deep sensory loss ranges from 30% to 50%, negatively impacting functional recovery (111). Proprioceptive impairment is associated with balance problems, gait disturbances, and an increased risk of falls (112).

Clinical Manifestations of Sensory Disorders: In chronic stroke, sensory impairments manifest in various ways. These disorders include hypesthesia (diminished sensation), paresthesia (abnormal sensation), decreased pain sensation, and decreased proprioceptive awareness. The location of the lesion also determines the type of sensory loss. For example, lesions to the thalamus or somatosensory cortex often cause severe superficial and deep sensory loss (113). These sensory impairments make it difficult for patients to recognize objects, coordinate their movements, and maintain balance. They negatively impact independence, particularly in activities of daily living, leading to a decrease in quality of life.

The Importance of the Sensory System in Rehabilitation: In chronic stroke rehabilitation, restoring sensory functions is as crucial as improving motor functions. The literature has shown that sensory stimulation and proprioceptive training programs have positive effects on improving motor functions (114). Stimulating the proprioceptive system promotes neuroplasticity, supports motor learning, and contributes to functional recovery. Furthermore, various studies have reported that closed kinetic chain exercises and sensory-based movement training are effective in strengthening the proprioceptive system (115). These exercises increase somatosensory input by stimulating joint and muscle receptors and improve balance and postural control. 4.13 Treatments for Knee Joint Sensation in Chronic Stroke

Decreased knee joint proprioception in chronic stroke patients is primarily due to two main factors: damage to somatosensory pathways in the central nervous system and inadequate stimulation of peripheral mechanoreceptors. Stroke damages the somatosensory cortex and brain regions responsible for processing sensory information from the joint, leading to impaired proprioceptive perception (114). Furthermore, post-stroke muscle tone changes, spasticity, and movement limitations reduce the stimulation of mechanoreceptors around the knee, leading to decreased sensory signals at the spinal and brainstem levels (116). In light of these pathological processes, the goal of chronic stroke rehabilitation is to reactivate and reorganize both central and peripheral sensory systems. The treatment methods used for this include:

Kinesio Taping Closed Kinetic Chain Exercises: Closed kinetic chain exercises involve moving the knee joint in functional positions, supporting the patient's body weight. These exercises activate muscle and joint receptors surrounding the knee, increasing stimulation of mechanoreceptors and enhancing proprioceptive input. Closed kinetic chain exercises have been shown to provide significant improvements in balance and proprioception in chronic stroke patients (115).

Manual Therapy and Joint Mobilizations: These techniques increase the sensitivity of mechanoreceptors through controlled movements applied to the knee joint capsule and surrounding tissues. This increases joint range of motion and supports proprioceptive perception. Manual therapy enhances peripheral sensory signals, enabling more effective input to the central nervous system (114,116).

Functional Electrical Stimulation: FES increases muscle activity through electrical stimulation of the muscles and stimulates sensory nerves surrounding the knee. This method supports both motor learning and improves sensory information flow. It has been reported that FES-assisted rehabilitation improves proprioceptive functions and walking performance in chronic stroke patients (117).

Virtual Reality (VR)-Based Rehabilitation: VR environments enhance sensory-motor integration by providing patients with real-time visual and auditory feedback. This supports brain plasticity and promotes restructuring in the somatosensory system. VR-assisted treatments have been shown to significantly improve lower extremity sensory functions and balance in chronic stroke patients (118).

Complementary Methods (Vibration Therapy and Neurofeedback): These methods aim to increase patients' sensory awareness. Vibration therapy provides direct stimulation of mechanoreceptors, while neurofeedback supports sensory-motor learning processes by facilitating patient control of their own neural activity (116).

In conclusion, decreased knee joint proprioception after chronic stroke is due to changes in both the central and peripheral nervous systems. Therefore, the rehabilitation process aims to reorganize the sensory and motor systems together by combining different treatment modalities.

4.13.1 Benefits of Closed Kinetic Chain Exercises Closed Kinetic Chain (CKC) exercises simultaneously target both stability and functionality through constant contact of the extremity with the support surface. One of the greatest advantages of these exercises is their potential to stimulate neuroplasticity by simultaneously activating cortical and subcortical areas due to their multi-joint movements (119). CKC exercises, especially for the lower extremities (e.g., squat, step-up, mini lunge), support the reactivation of weakened muscles on the hemiplegic side while also strengthening sensorimotor integration.Thus, both muscle strength and muscle control are improved (120). Research has shown that CKC exercises reduce asymmetrical posture patterns in post-stroke patients, balance weight transfer, and increase gait symmetry (121). Kang and Kim (2013) reported significant improvements in static and dynamic balance skills in stroke patients who underwent CKC exercises (120). CKC exercises also improve lower extremity positional perception by increasing proprioceptive feedback. Knee joint proprioception, which is frequently impaired after stroke, can be restored through closed-chain exercises, particularly in weight-bearing positions (115). This directly contributes to reducing the risk of falls and promoting safe mobility. Another study found significant improvements in objective measures such as the Fugl-Meyer Motor Score, the Timed Up and Go test, and the Berg Balance Scale in individuals who underwent CKC exercises.

KC exercises also increase patient motivation and participation in rehabilitation thanks to their focus on functional goals, reducing secondary complications related to fatigue and inactivity. Furthermore, these exercises, which integrate sensorimotor and cognitive inputs, provide broader neurological benefits by affecting both upper and lower motor neuron systems (122). Consequently, closed kinetic chain exercises not only increase muscle strength, but also strengthen proprioception, improve balance, functionally improve gait, and support recovery in the central nervous system, providing a multidimensional contribution to the post-stroke rehabilitation process.

4.13.2 Benefits of Kinesiotaping Kinesiotaping is a treatment method that uses flexible, elastic tape applied to the skin and aims to have multiple effects on the musculoskeletal and nervous systems. Considering the motor deficits, tone imbalances, proprioceptive deficits, and functional disabilities that occur after stroke, kinesio taping stands out as a supportive rehabilitation modality, especially in the chronic phase (11).

One of the most common problems in individuals with chronic stroke is imbalance resulting from muscle weakness and increased tone on the hemiplegic side. Kinesio taping stimulates mechanoreceptors on the skin in the applied area, increasing proprioceptive feedback and helping to normalize muscle activity. The basis of this effect is the activation of nerve endings by the micro-tension created by the tape on the skin, thus increasing the sensory impulse sent to the central nervous system (12).

Recent studies have reported that kinesiotaping leads to significant improvements in areas such as posture control, balance, walking speed, and pain management in chronic stroke patients. Kinesiotaping applied around the knee has been shown to improve static and dynamic balance in hemiplegic individuals (123). Application of taping on the ankle has been reported to improve gait symmetry and standing time (124). Another recent study found that kinesiotaping applied to individuals experiencing shoulder subluxation after stroke reduced pain and improved functional range of motion by increasing shoulder stability (125). These results demonstrate that the support and postural correction effects it provides to the musculoskeletal system are not limited to the lower extremities. Furthermore, the application of kinesiotaping in conjunction with conventional physiotherapy leads to more significant functional improvements. It is emphasized that it opens up new possibilities. Comparative studies have reported that when taping is added to exercise programs, higher Berg Balance Score, Timed Up and Go time, and 10-Meter Walk Test scores are achieved compared to groups receiving exercise alone (123).

Kinesio taping is an effective complementary approach in chronic stroke rehabilitation because it is non-invasive, easy to apply, cost-effective, and has high patient compliance. However, application techniques based on accurate anatomical knowledge and tailoring to the individual patient profile are decisive factors in its effectiveness.

4.14 Assessment of Knee Joint Sensation Knee joint sensation is a fundamental component of motor control, particularly in terms of proprioception, movement, and position perception. Impairments in knee joint sensation can occur in chronic stroke, orthopedic injuries, and other neurological conditions. Therefore, accurate and systematic assessment of knee joint sensation is important for treatment planning and monitoring the rehabilitation process. Passive and Active Position Sense Tests (Joint Position Sense - JPS): The knee is moved passively or actively at certain angles. The patient is asked to estimate the position of the knee. Proprioception is evaluated by measuring the accuracy of position perception. (126)Motion Detection Threshold Test (TTDPM): Passive movement of the knee is initiated at very small angles. The patient's time to detect movement and sensitivity are recorded. (127) Vibration Sense Tests: Vibration is applied to the relevant area of the knee. Vibration perception ability is assessed and nerve and proprioceptive function is measured. (128) Functional Tests Berg Balance Scale (BBS): Measures static and dynamic balance performance. Time Up and Go (TUG) Test: Assesses functional mobility. Balance Platform and Gait Analysis: Dynamic balance and gait symmetry measurements are performed.

1.5. Electrophysiological Tests: Contributes to the assessment of proprioceptive functions by measuring nerve conduction velocity and reflex responses.

Evaluation of knee joint sensation with objective and functional measurements is critical for monitoring treatment effectiveness and for personalized rehabilitation planning. Proprioceptive losses are closely related to balance disorders and walking problems; Therefore, early and accurate evaluation is necessary for functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a stroke more than 6 months ago,
* Individuals with a medically stable condition,
* Ability to understand simple instructions,
* Individuals with spasticity graded between 0 and 2 according to the Modified Ashworth Scale,
* Individuals who can walk independently or with assistive devices,
* Individuals who agree to participate in the study and are able to comply with the study procedures.

Exclusion Criteria:

* Severe cognitive impairment (Mini-Mental Test score < 24),
* Orthopedic conditions that may cause knee pain during exercise,
* Other neurological conditions that may affect proprioception,
* Severe joint contracture,
* Individuals who do not wish to voluntarily participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of knee joint position sense | 2 months
  Knee joint position sense will be evaluated using active and passive joint position sense tests. Prior to testing, the limb will be passively moved 10 times to prepare for the movement. The Physiomaster mobile application will be used to measure the angular difference between the affected and unaffected knees at the end of the movement.
  Active joint position sense will be measured by asking participants to replicate a 45° knee flexion angle with their eyes closed. The angular error will be calculated.
  Passive joint position sense will be assessed by passively positioning the knee, then asking participants to estimate the angle after returning to the starting position. Repetitive flexion and extension movements will be performed, and error detection will be recorded. Placebo movements will be included in the evaluation.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | 2 months
  The Berg Balance Scale (BBS) is used to assess individuals' static and dynamic balance.
  It consists of 14 items that evaluate the ability to maintain balance during various positions, postural changes, and movements. The assessment is based on the individual's ability to perform each task either independently or within a specific time or distance.
  Each item is scored on a scale from 0 to 4, where 0 indicates inability to perform the task, and 4 reflects normal performance.
  The maximum total score is 56.
  * A score between 0-20 suggests that the individual is dependent on a wheelchair and has a 100% risk of falling.
  * A score between 21-40 indicates that the person is at risk of falling and may require assistance for walking.
  * A score between 41-56 implies that the individual can ambulate independently with minimal fall risk.
Timed Up and Go Test (TUG) | 2 months
  The Timed Up and Go Test (TUG) is used to assess functional mobility. In the TUG test, the time it takes for the participant to stand up from a chair, walk 3 meters, turn around, walk back, and sit down again will be measured.
10-Meter Walk Test (10MWT) | 2 months
  The 10-Meter Walk Test (10MWT) is used to determine walking speed. Participants will perform 2-3 trials at both their self-selected comfortable speed and maximum safe speed. Instructions will be given to walk either at a "normal, comfortable pace" or "as fast as possible in a safe manner."
  No practice trials will be conducted, and participants will be allowed to rest for at least 30 seconds between trials. Typical footwear, usual orthoses, and necessary assistive devices will be used during testing.
  Participants will walk approximately 14 meters, which includes a 2-meter acceleration zone, a 6-meter timed middle section, and a 2-meter deceleration zone. The time to walk the middle 6 meters will be recorded using a stopwatch, starting when the participant's toe crosses the starting cone and stopping when the toe crosses the ending cone.
  Walking speed will be calculated for each trial.
Stroke-Specific Quality of Life Scale (SS-QOL) | 2 months
  Quality of life is also an important prognostic indicator in stroke and allows for a broader understanding of the disease.
  The Stroke-Specific Quality of Life Scale (SS-QOL) consists of 49 items across 12 domains: mobility, energy, upper extremity function, work/productivity, mood, self-care, social roles, family roles, vision, language, thinking, and personality.
  The SS-QOL items are rated using a 5-point Likert scale, with responses ranging from 1 (Strongly disagree) to 5 (Strongly agree).
  Higher scores on the scale indicate a better quality of life, while lower scores reflect a poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dilanur Ö Özkaraoğlu, Doctor Physiotherapist, Study Director — Medipol University
Locations (1):
- Özel İncirli Akademi Özel eğitim ve rehabilitasyon merkezi, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study has not yet been completed. All data collected will be used solely for purposes approved by the ethics committee and will not be shared with third parties. Since no specific consent was obtained from participants for IPD sharing, data will not be shared in accordance with confidentiality and ethical principles.